CLINICAL TRIAL: NCT03379038
Title: Role Of Physical Therapy In Relieving Constipation In Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Waqar Ahmed Awan, Assistant Professor, Isra University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IIRS-IUISB/PHD/007
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2017-12

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Spasticity; Constipation; Gross Motor Functional Classification Scale; Defecation Frequency; Constipation Severity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Constipation

STUDY DESIGN:
Intervention Model Description: The two groups were progressive physical therapy group and maintenance physical therapy group. For any given subject, spasticity, defecation frequency and constipation severity evaluations were completed on the same day. Each subject in PPT group completed 6 weeks of physical therapy sessions which were aimed to decrease spasticity, increase ROM, and improve strength and functional activity level. Each subject was evaluated for changes in symptoms on, 2nd week, 4th week and 6th week. In MPT group same protocol was used but the aim was to maintain current status of level of spasticity, ROM, strength and functional activity. After 6 weeks of physical therapy sessions were completed both groups underwent a 2-week washout period to eliminate the effects of 6-week physical therapy. After the washout period subjects were crossed over from PPT group to MPT group and vice versa.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Physical Therapy (PPT) (Experimental): Duration: Each child was given 40-minute session. Frequency: Two sets were performed, 5-10 active assisted sit-ups in each set at least once a day. Furthermore, the subjects were advised to use CP chair and standing frame/wall corner for sitting/standing position respectively for at least 15-30 minutes once a day. These exercises were followed by reflex inhibiting postures in sitting and lying positions.
  Total 42 sessions were performed in 6 weeks (7 days/week). Intensity: The aim of the PPT was to improve the patient's level of spasticity, strength and activity level.
  Interventions: Other: Progressive Physical Therapy
- Maintenance Physical Therapy (MPT) (Placebo Comparator): Duration: Each child was given 40-minute session. Frequency: Two sets were performed, 5-10 active assisted sit-ups in each set at least once a day. Furthermore, the subjects were advised to use CP chair and standing frame/wall corner for sitting/standing position respectively for at least 15-30 minutes once a day. These exercises were followed by reflex inhibiting postures in sitting and lying positions. Total 42 sessions were performed in 6 weeks (7 days/week).
  Intensity:The aim of the MPT was to maintain the patient's current level of spasticity, strength and activity level.
  Interventions: Other: Maintenance Physical Therapy

INTERVENTIONS:
Other: Progressive Physical Therapy — Stretching of the tight muscle, positioning, abdominal co activation; rolling etc to decrease muscle tone and functional independence.
  Arms: Progressive Physical Therapy (PPT)
Other: Maintenance Physical Therapy — Same Physical therapy protocol but aim was to maintain current level of spasticity and functioning
  Arms: Maintenance Physical Therapy (MPT)

SUMMARY:
This study was conducted to determine the effectiveness of Physical Therapy management in relieving constipation among Spastic Cerebral Palsy children. There were two groups, Group A received routine Physical Therapy and Group B received maintenance Physical Therapy (aim to maintain current level of spasticity, functionality to avoid deterioration of conadition as approved by ASRC)

DETAILED DESCRIPTION:
Physical therapy makes an integral part of the non-pharmacological, conservative management of cerebral palsy. Routine physical therapy aims to reduce spasticity, improve joint range of motion (ROM), and improve strength and mobility.

Passive ROM and stretching of lower limb and trunk increases parasympathetic activity and thus improves intestinal motility in prolonged bed ridden patients.Abdominal muscle training improves intestinal motility by two ways: mechanically by improving fecal propulsion towards rectum and neurologically by inducing parasympathetic activity to improve intestinal motility.20 Thermotherapy of back and abdomen in chronic constipation patient improves intestinal blood flow and parasympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the recruitment in the study were: spastic CP children on oral feeding with constipation between ages 2-12 years of both genders, spasticity above 1+ grade on modified Ashworth scale, functional activity level between 2-5 grades on gross motor functional classification scale (GMFCS).

Exclusion Criteria:

* CP children with other systemic co-morbidities, physical deformity in GIT and intellectual disability were excluded from the study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Spastcity Spasticity | 6 Weeks
  Modified Ashworth scale (MAS)
  * 0 = No increase in muscle tone
  * 1 = Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  * 1+ = Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  * 2 = More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  * 3 = Considerable increase in muscle tone, passive movement difficult.
  * 4 = Affected part(s) rigid in flexion or extension
Defecation Frequency (DF) | 6 weeks
  Defecation frequency less than three times a week was considered constipation and measured by nominal scale 1= twice a month, 2= once a week, 3= twice a week and 4= daily
Constipation assessment scale (CAS) | 6 Weeks
  used to determine the severity of constipation. The CAS consists of eight characteristics. Each of these characteristics is given a three point rating scale (0= no problem, 1= some problem, 2= severe problem). These scores are summed up to make a range from 0 for no constipation to 16 for the most severe constipation

CONTACTS AND LOCATIONS:
Locations (1):
- Isra Institute or Rehabilitation Sciences, Isra University Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR